CLINICAL TRIAL: NCT01021774
Title: Comparison of Anal Fistula Treatment Outcome - Collagen Plug vs Advancement Flap Surgery. A Randomised Prospective Blinded Multi-centre Study
Brief Title: Anal Fistula Treatment Outcome - Collagen Plug Versus Advancement Flap Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Uppsala University Hospital (Other); University Hospital, Linkoeping (Other); Region Örebro County (Other)
Responsible Party: Principal Investigator, Tom Oresland, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-08493(REK)
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Perianal Fistula
MeSH Terms: interventions — Portacaval Shunt, Surgical; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advancement flap surgery (Active Comparator)
  Interventions: Procedure: Anal fistula treatment
- Collagen plug (Active Comparator)
  Interventions: Procedure: Anal fistula treatment

INTERVENTIONS:
Procedure: Anal fistula treatment — A comparison of collagen plug vs advancement flap surgery
  Other Names: Perianal; Lambeau technique; Anal fistula plug; Fistula; Surgical treatment

SUMMARY:
The purpose of this study is to determine whether the outcome of anal fistula repair with a collagen plug is comparable to that of repair by a mucosal advancement flap.

DETAILED DESCRIPTION:
Perianal fistula can occur as a complication to a perianal abscess. A perianal fistula is associated with significant morbidity and reduced quality of life. Anal fistulas seldom heal spontaneously and may require surgical intervention. The main purpose of the operation will be to close the fistula and preserve anal continence. The traditional surgical fistula closing techniques often show disappointing results. Today, a collagen plug for fistula treatment is commercially available. The mounting of this plug is technically easy and less invasive than the traditional closure of the fistula by making a lid of anal mucosa (advancement flap). The purpose of this study is to determine whether the outcome of anal fistula repair with a collagen plug is comparable to that of repair by a mucosal advancement flap, with regard to healing of fistula, anal continence and pain. Plug treatment has so far shown promising results, but prospective, randomised controlled trials are needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fistula involving > 1/3 of the external anal sphincter
* Single, continuous fistula tract at time of inclusion (implies pre-treatment with seton)
* Patients with previous fistula surgery can be included (max. 1 lambeau or 1 plug)
* All patients included must be able to fill in an informed, written consent and to understand its implications and contents and to participate in the follow-up

Exclusion Criteria:

* Fistula tract shorter than 2 cm
* Complex fistula tract system (branching of the fistula tract)
* Age < 18 years
* Pregnancy
* HIV-positivity
* Fistula caused by malignancy
* Tuberculosis
* Hidrosadenitis suppurativa
* Pilonidal sinus disease
* No internal fistula opening found
* Unable/contra indications to go through MRI scanning
* Crohn´s disease
* Ulcerative proctitis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-11; Primary Completion 2015-07 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Anorectal fistula closing rate | 1 year

SECONDARY OUTCOMES:
Quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tom Oresland, M.D., Ph.D., Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lorenskog, Norway

REFERENCES:
- [Derived] Bondi J, Avdagic J, Karlbom U, Hallbook O, Kalman D, Saltyte Benth J, Naimy N, Oresland T. Randomized clinical trial comparing collagen plug and advancement flap for trans-sphincteric anal fistula. Br J Surg. 2017 Aug;104(9):1160-1166. doi: 10.1002/bjs.10549. Epub 2017 May 10. PMID 28489253